CLINICAL TRIAL: NCT02623426
Title: Macular Edema Ranibizumab v. Intravitreal Anti-inflammatory Therapy Trial
Acronym: MERIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 119247; U10EY024527 (NIH); ML29257 (Other: Genentech (donating ranibizumab for US clinics)
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Uveitis; Macular Edema
Keywords: uveitic macular edema; uveitis
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — Dexamethasone; Calcium Dobesilate; Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dexamethasone intravitreal implant 0.7mg (Active Comparator): Participants were randomized to a treatment group. A participant may have 1 or 2 eyes with macular edema (eligible eyes) receiving the same treatment.
  Eligible eye(s) treated at study visit M01 (week 0).
  Retreatment required at study visit M03 (8 weeks) if re-treatment criteria met.
  Retreatment permitted at later time points if retreatment criteria met.
  Re-treatment criteria:
  1. Central subfield thickness greater than 1.1X upper limit of normal (330 μm for Zeiss and Topcon Spectral Domain (SD) Optical Coherence Tomography (OCT) and 352 μm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted)
  Minimum time between treatments: minimum target is 8 weeks after last injection but re-injection permitted as early as 51 days after last injection;
  Interventions: Drug: Dexamethasone intravitreal implant 0.7 mg
- Intravitreal methotrexate 400µg in 0.1mL (Active Comparator): Participants were randomized to a treatment group. A participant may have 1 or 2 eyes with macular edema (eligible eyes) receiving the same treatment.
  Eligible eye(s) treated at study visit M01 (week 0).
  Retreatment required at M02 (4 weeks) and M03 (8 weeks) if retreatment criteria met.
  Retreatment permitted at later time points if retreatment criteria met.
  Minimum time between treatments: minimum target is 4 weeks after last injection but re-injection permitted as early as 23 days after last injection.
  Interventions: Drug: Intravitreal Methotrexate 400 µg
- Intravitreal ranibizumab 0.5mg in 0.05mL (Active Comparator): Participants were randomized to a treatment group. A participant may have 1 or 2 eyes with macular edema (eligible eyes) receiving the same treatment.
  Eligible eye(s) treated at study visits M01 (week 0), M02 (4 weeks), and M03 (8 weeks).
  Retreatment permitted at M04 (12 weeks) and at later time points if retreatment criteria met.
  Minimum time between treatments: minimum target is 4 weeks after last injection but re-injection permitted as early as 23 days after last injection.
  Re-treatment permitted at later time points if re-treatment criteria met.
  Interventions: Drug: Intravitreal Ranibizumab 0.5 mg

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant 0.7 mg — Standard preparation as described for intravitreal injections.
  Other Names: Ozurdex
  Arms: Dexamethasone intravitreal implant 0.7mg
Drug: Intravitreal Methotrexate 400 µg — Intravitreal Methotrexate 400 µg injection procedures should be carried out under controlled aseptic conditions which include the use of sterile gloves and a sterile eyelid speculum (or equivalent). Adequate anesthesia and a broad-spectrum microbicide such as betadine, applied to the periocular skin, eyelid and ocular surface are required prior to the injection.
  Arms: Intravitreal methotrexate 400µg in 0.1mL
Drug: Intravitreal Ranibizumab 0.5 mg — Intravitreal Ranibizumab 0.5 mg injection procedures should be carried out under controlled aseptic conditions which include the use of sterile gloves and a sterile eyelid speculum (or equivalent). Adequate anesthesia and a broad-spectrum microbicide such as betadine, applied to the periocular skin, eyelid and ocular surface are required prior to the injection.
  Other Names: Lucentis
  Arms: Intravitreal ranibizumab 0.5mg in 0.05mL

SUMMARY:
The Macular Edema Ranibizumab v. Intravitreal anti-inflammatory Therapy (MERIT) Trial will compare the relative efficacy and safety of intravitreal methotrexate, intravitreal ranibizumab, and the intravitreal dexamethasone implant for the treatment of uveitic macular edema persisting or reoccurring after an intravitreal corticosteroid injection. MERIT is a parallel design (1:1:1), randomized comparative trial with an anniversary close-out after 6 months of follow-up. The primary outcome is percent change in central subfield thickness from the baseline OCT measurement to the 12 week visit.

DETAILED DESCRIPTION:
Macular edema (ME) is the most common structural complication and cause of visual impairment and legal blindness in uveitis patients. Traditional approaches to the treatment of uveitic ME have included the use of regional corticosteroid therapy, delivered periocularly, including posterior sub-Tenon's and orbital floor injections, or via the intravitreal route. While corticosteroid injections may reduce ME and improve vision, the effect is often variable with a limited duration. Persistent macular edema is a common occurrence and often requires repeated intravitreal injections of corticosteroids, which expose eyes to a significant risk of increased intraocular pressure ocular and cataract development. The often refractory nature of uveitic ME and its impact on visual function underscores the need to identify effective alternative medical therapeutic options. Recent pilot studies have shown intravitreal methotrexate (MTX) and intravitreal ranibizumab (Lucentis®, Genentech Inc., San Francisco, CA) to be promising treatments for uveitic ME, and intravitreal dexamethasone implant (Ozurdex®, Allergan, Irvine, CA) has recently been approved by the U.S. FDA for uveitic ME in patients with non-infectious uveitis. In addition to being effective, intravitreal MTX and ranibizumab potentially may have less ocular side effects than corticosteroids, particularly less IOP elevation. However, the relative efficacy of these treatments is unknown. The Macular Edema Ranibizumab v. Intravitreal anti-inflammatory Therapy (MERIT) Trial will compare the relative efficacy and safety of intravitreal methotrexate, ranibizumab, and dexamethasone implant. MERIT is a parallel design (1:1:1), randomized comparative effectiveness trial with an anniversary close-out after 6 months of follow-up. The primary outcome is percent change in central subfield thickness from the baseline OCT measurement to the 12 week visit.

ELIGIBILITY:
Inclusion criteria:

Patient level inclusion criterion

1. 18 years of age or older;

   Eye level inclusion criteria - at least one eye must meet all of the following conditions
2. Inactive or minimally active non-infectious anterior, intermediate, posterior or panuveitis, as defined by the Standardization of Uveitis Nomenclature (SUN) Working Group criteria as ≤ 0.5+ anterior chamber cells, ≤ 0.5+ vitreous haze grade and no active retinal/choroidal lesions for a minimum of 4 weeks;
3. Macular edema (ME) defined as the presence of macular thickness greater than the normal range for the OCT machine being used (see cut points below), regardless of the presence of cysts, following an intravitreal corticosteroid injection (≥ 4 weeks following intravitreal triamcinolone injection or ≥ 12 weeks following intravitreal dexamethasone implant injection);

   Greater than 300 μm for Zeiss Cirrus Greater than 320 μm for Heidelberg Spectralis Greater than 300 μm for Topcon SD OCT
4. Baseline fluorescein angiogram that, as assessed by the study ophthalmologist, is gradable for degree of leakage in the central subfield;
5. Best corrected visual acuity (BCVA) 5/200 or better;
6. Baseline intraocular pressure > 5 mm Hg and ≤ 21 mm Hg (current use of ≤3 intraocular pressure-lowering medications and/or prior glaucoma surgery are acceptable (Note: combination medications, e.g., Combigan, are counted as two IOP-lowering medications);
7. Media clarity and pupillary dilation sufficient to allow OCT testing and assessment of the fundus.

Exclusion criteria:

Patient level exclusion criteria

1. History of infectious uveitis in either eye;
2. History of infectious scleritis of any type in either eye (Note: History of noninfectious scleritis that has been active in past 12 months is an eye-level exclusion -see #13 below);
3. History of keratitis (with the exception of keratitis due to dry eye) in either eye;
4. History of central serous retinopathy in either eye;
5. Active infectious conjunctivitis in either eye;
6. Oral prednisone dose > 10 mg per day (or of an alternative corticosteroid at a dose higher than that equipotent to prednisone 10 mg per day) OR oral prednisone dose ≤ 10 mg per day at baseline that has not been stable for at least 4 weeks (note: if patient is off of oral prednisone at baseline (M01 study visit) dose stability requirement for past 4 weeks does not apply);
7. Systemic immunosuppressive drug therapy that has not been stable for at least 4 weeks (note: use of systemic methotrexate is acceptable as long as regimen has been stable for at least 4 weeks);
8. Use of oral acetazolamide or other systemic carbonic anhydrase inhibitor at baseline;
9. Known allergy or hypersensitivity to any component of the study drugs;
10. For women of childbearing potential: pregnancy, breastfeeding, or a positive pregnancy test; unwilling to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for duration of trial;

    Eye level exclusion criteria - at least one eye that meets all inclusion criteria cannot have any of the following conditions
11. History of infectious endophthalmitis;
12. History of severe glaucoma as defined by optic nerve damage (cup/disc ratio of ≥ 0.9 or any notching of optic nerve to the rim);
13. History of active noninfectious scleritis in past 12 months (Note: History of noninfectious scleritis is acceptable if the last episode of active scleritis resolved at least 12 months prior to enrollment);
14. Presence of an epiretinal membrane noted clinically or by OCT that per the judgment of study ophthalmologist may be significant enough to limit improvement of ME (i.e., causing substantial wrinkling of the retinal surface);
15. Torn or ruptured posterior lens capsule
16. Presence of silicone oil;
17. Ozurdex administered in past 12 weeks;
18. Anti-vascular endothelial growth factor (VEGF) agent, intravitreal methotrexate, or intravitreal/periocular corticosteroid administered in past 4 weeks;
19. Fluocinolone acetonide implant (Retisert) placed in past 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Jabs, MD, MBA, Study Chair — Center for Clinical Trials and Evidence Synthesis, JHU, Baltimore, MD
Locations (33):
- United States (19):
  - Jules Stein Eye Institute, UCLA, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Anne Bates Leach Eye Hospital, University of Miami Miller School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Duke Eye Center, Duke University, Durham, North Carolina
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
  - MidAtlanitc Retina, Wills Eye Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt, Nashville, Tennessee
  - Retinal Consultants of Houston, Houston, Texas
  - John A. Moran Eye Center, University of Utah, Salt Lake City, Utah
- Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria, Australia
- McGill University, Montreal, Quebec, Canada
- India (4):
  - LV Prasad Eye Institute - Bhubaneswar, Bhubaneswar, Odisha
  - Medical and Vision Research Foundation, Chennai, Tamil Nadu
  - LV Prasad Eye Institute - Hyderabad, Hyderabad, Telangana
  - Advanced Eye Center, Post Graduate Institute of Medical Education and Research, Chandigarh
- United Kingdom (8):
  - University Hospitals Bristol NHS Foundation Trust, Bristol, England
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - University Hospitals of Leicester NHS Trust, Leicester, England
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool, England
  - Moorfields Eye Hospital NHS Foundation Trust, London, England
  - Manchester University NHS Foundation Trust, Manchester, England
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Moorfields Eye Hospital, London

REFERENCES:
- [Derived] Multicenter Uveitis Steroid Treatment Trial (MUST) Research Group, Writing Committee:; Acharya NR, Vitale AT, Sugar EA, Holbrook JT, Burke AE, Thorne JE, Altaweel MM, Kempen JH, Jabs DA. Intravitreal Therapy for Uveitic Macular Edema-Ranibizumab versus Methotrexate versus the Dexamethasone Implant: The MERIT Trial Results. Ophthalmology. 2023 Sep;130(9):914-923. doi: 10.1016/j.ophtha.2023.04.011. Epub 2023 Jun 13. PMID 37318415

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection: Participants were randomized to a treatment group. A participant may have 1 or 2 eyes with macular edema receiving the same treatment.
  Ozurdex (0.7 mg dexamethasone pellet) delivered via intravitreal injection at week 0 Second injection required at Week 8 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria is met.
  Retreatment criteria :
  1. Central subfield thickness greater than 1.1 times the upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
- Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free: Participants were randomized to a treatment group. A participant may have 1 or 2 eyes with macular edema receiving the same treatment. Intravitreal methotrexate 400 µg in 0.1 mL Eligible eye(s) treated M01+ Retreatment required at M02, M03 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria met
  Retreatment criteria:
  1. Central subfield thickness greater than 1.1 times the upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
- Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL: Participants were randomized to a treatment group. A participant may have 1 or 2 eyes with macular edema receiving the same treatment. Intravitreal ranibizumab (Lucentis) 0.5 mg in 0.05 mL Eligible eye(s) treated M01+ Retreatment required at M02, M03 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria met
  Retreatment criteria:
  1) Central subfield thickness greater than 1.1 times the upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
Period: Overall Study
Arm/Group | Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection | Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free | Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL
Started | 65; 77 eyes | 65; 79 eyes | 64; 69 eyes
4 Week Visit | 65; 77 eyes | 64; 78 eyes | 63; 68 eyes
8 Week Visit | 65; 77 eyes | 64; 78 eyes | 61; 66 eyes
Completed (12 week visit) | 64; 76 eyes | 63; 77 eyes | 61; 66 eyes
Not Completed | 1; 1 eyes | 2; 2 eyes | 3; 3 eyes
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Randomized participants had 1 or both eyes with macular edema, defined as the presence of central subfield macular thickness greater than the normal range for the OCT machine being used
Units Other Than Participants: Eyes with Macular Edema
Groups:
- Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection: Ozurdex (0.7 mg dexamethasone pellet) delivered via intravitreal injection at week 0 Eligible eye (s) treated at week 0 Second injection required at Week 8 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria is met.
  Retreatment criteria :
  1. Central subfield thickness greater than 1.1 times upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
- Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free: Intravitreal methotrexate 400 µg in 0.1 mL Eligible eye(s) treated at week 0 Retreatment required at M02, M03 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria met
  Retreatment criteria:
  1. Central subfield thickness greater than 1.1 times upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
- Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL: Intravitreal ranibizumab (Lucentis) 0.5 mg in 0.05 mL Eligible eye(s) treated M01+ Retreatment required at M02, M03 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria met
  Retreatment criteria:
  1) Central subfield thickness greater than 1.1 times upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
- Total: Total of all reporting groups
Arm/Group | Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection | Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free | Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL | Total
Number analyzed (Participants) | 65 | 65 | 64 | 194
Number analyzed (Eyes with Macular Edema) | 77 | 79 | 69 | 225
Age, Continuous [Median (Full Range); unit: years] | 59 [18 to 81] | 59 [20 to 83] | 57 [24 to 83] | 58 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 40 | 129
  Male | 24 | 17 | 24 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 64 | 63 | 62 | 189
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 8 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 22 | 13 | 51
  White | 38 | 28 | 41 | 107
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 2 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 1 | 8
  United States | 40 | 43 | 44 | 127
  United Kingdom | 9 | 8 | 8 | 25
  Australia | 2 | 2 | 3 | 7
  India | 10 | 9 | 8 | 27
Intraocular pressure (IOP) [Median (Full Range); unit: mm Hg] — Population: Eyes with macular edema
  mm Hg | 15 [5 to 21] | 15 [5 to 23] | 14 [7 to 21] | 14 [5 to 23]
Visual acuity [Median (Full Range); unit: Standard letters] — Measure Description: Participants' visual acuity was measured by certified examiners with best refractive correction in place. Participants were challenged with reading letters on lines of the standard ETDRS eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until no more meaningful readings could be made and were scored by how many letters could be correctly identified. More letters read is associated with higher visual acuity. (85 standard letters = 20/20 vision)
  Standard letters | 68 [25 to 89] | 64 [6 to 85] | 67 [6 to 88] | 66 [6 to 88]
Retinal thickness at the center subfield [Median (Full Range); unit: um] — Central subfield thickness as measured by OCT at a fundus photograph reading center
  um | 457 [241 to 1116] | 476 [276 to 991] | 401 [220 to 1091] | 453 [210 to 1116]
Concomitant systemic medication [Count of Participants; unit: Participants] — Count of participants on systemic medication for the treatment of macular edema or uveitis at the baseline visit
  Participants | 28 | 27 | 29 | 84

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Baseline Central Subfield Thickness Observed at 12 Weeks
Description: The primary outcome is the change in central subfield thickness from baseline to 12 weeks measured on a relative scale as the the proportion of the baseline central subfield thickness. The proportion of baseline subfield thickness is estimated by a mixed effect model that includes time points for baseline, week 4, week 8, and week 12 and the treatment group. The treatment effect is the interaction (product) of time point and treatment. Contrasts of the model parameter estimates were used to calculate the change from baseline to week 12 and the comparison between treatment groups.
  Values less than 1 indicate a decrease in retinal thickness with lower values indicating greater decreases (improvement).The OCT outcomes were measured by masked readers. The 12-week visit was chosen as the time to assess the primary outcome because of the ranibizumab treatment schedule and the peak effect time for dexamethasone
Time Frame: At 12-week visit
Measure: Mean (95% Confidence Interval); unit: Proportion of baseline retinal thickness
Units Other Than Participants: Eyes with macular edema
Groups:
- Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection: Ozurdex (0.7 mg dexamethasone pellet) delivered via intravitreal injection at week 0 Eligible eye (s) treated at week 0 Second injection required at Week 8 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria is met.
  Retreatment criteria :
  1. Central subfield thickness greater than 1.1 times the upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
- Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free: Intravitreal methotrexate 400 µg in 0.1 mL Eligible eye(s) treated at week 0 Retreatment required at M02, M03 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria met
  Retreatment criteria:
  1. Central subfield thickness greater than 1.1 times the upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
Arm/Group | Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection | Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free | Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL
Number analyzed (Participants) | 65 | 66 | 64
Number analyzed (Eyes with macular edema) | 77 | 79 | 69
Proportion of baseline retinal thickness | 0.65 [0.58 to 0.72] | 0.88 [0.81 to 0.96] | 0.79 [0.70 to 0.89]
Statistical Analysis 1: Comparison: Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection vs Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free; A sample size of 240 was calculated to provide 91% power to detect a 25% reduction for Ozurdex, a 38% reduction for Methotrexate and Lucentis assuming a standard deviation of 0.33, 25% with bilateral disease, between-eye correlation of 0.4, 10% loss to follow-up, and a two-sided type 1 error rate of 0.025 for each pairwise comparison; Test type: Superiority; p < 0.001, mixed effects model — A Bonferroni correction was used to adjust for the co-primary hypotheses;a two-sided type I error rate of 0.05/2 = 0.025 was used to determine statistical significance for the two pairwise comparisons (Ozurdex vs Methotrexate and Ozurdex vs Lucentis); Ratio of the proportion of baseline = 1.36, 95% CI 2-sided [1.19 to 1.56] — The treatment effect is the ratio of the proportions of baseline retinal thickness (Methotrexate/Ozurdex). Values greater than 1 indicate less reduction in retinal thickness in the Methotrexate treated group compared to Ozurdex
Statistical Analysis 2: Comparison: Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection vs Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.012, mixed effects model — [p-value comment as in outcome 1, analysis 1]; Ratio of the proportion of BL = 1.22, 95% CI 2-sided [1.04 to 1.43] — The treatment effect is the ratio of the proportions of baseline retinal thickness (Lucentis/Ozurdex) at 12 weeks. Values greater than 1 indicate less reduction in retinal thickness in the Lucentis treated group compared to Ozurdex

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Serious adverse events were reported via an expediated reporting system followed by medical safety review. Non-serious events were collected by non-systemic means via an adverse event log that was completed at each visit and by systemic collection of information on ocular events of special interest on the follow up visit case reform forms.
Groups:
- Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection: Ozurdex (0.7 mg dexamethasone pellet) delivered via intravitreal injection at week 0 Eligible eye (s) treated at week 0 Second injection required at Week 8 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria is met.
  Retreatment criteria :
  1. Central subfield thickness greater than 1.1X upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
- Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free: Intravitreal methotrexate 400 µg in 0.1 mL Eligible eye(s) treated at week 0 Retreatment required at M02, M03 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria met
  Retreatment criteria:
  1. Central subfield thickness greater than 1.1X upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
  2. IOP of <25 mm Hg (treatment with ≤3 IOP-lowering agents permitted), IOP criteria for initial injection of study treatment in eligible eye(s) is ≤21 mm Hg with ≤3 IOP-lowering agents
- Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL: Intravitreal ranibizumab (Lucentis) 0.5 mg in 0.05 mL Eligible eye(s) treated M01+ Retreatment required at M02, M03 if retreatment criteria met Retreatment permitted at M04 and later if retreatment criteria met
  Retreatment criteria:
  1) Central subfield thickness greater than 1.1X upper limit of normal (330 µm for Zeiss and Topcon SD OCT and 352 µm for Heidelberg OCT) and/or cystoid space(s) within 1 mm central subfield.
Arm/Group | Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection | Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free | Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/64
Serious Adverse Events (participants affected / at risk) | 6/65 | 7/65 | 3/64
Other Adverse Events (participants affected / at risk) | 12/65 | 24/65 | 14/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection (N=65) | Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free (N=65) | Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL (N=64)
glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure decreased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Eye disorders) | 3 (4) | 0 (0) | 0 (0)
Iridotomy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual acuity decreased (Eye disorders) | 0 (0) | 4 (4) | 1 (1) — Decrease from baseline of >= 30 standard letters (6 lines on eye chart)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Catheterization cardiac for hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vasovagal response (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex (0.7 mg Dexamethasone Pellet) Delivered Via Intravitreal Injection (N=65) | Intravitreal Methotrexate 400 µg in 0.1 mL 0.9% Sodium Chloride Solution, Preservative-free (N=65) | Intravitreal Ranibizumab (Lucentis) 0.5 mg in 0.05 mL (N=64)
Eye pain (Eye disorders) | 5 (7) | 5 (7) | 4 (5)
Ocular hypertension (Eye disorders) | 3 (3) | 2 (2) | 1 (1)
Uveitis (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Vitreous or subconjunctival hemorrhage (Eye disorders) | 3 (3) | 0 (0) | 1 (1) — Systemic collection on case report form
Surgery to control IOP (Eye disorders) | 1 (1) | 4 (4) | 0 (0) — Systemic collection on case report form of surgery to control IOP (e.g. tube/shunt, paracentesis)
Post injection IOP increase >=30 mmHg (General disorders) | 0 (0) | 12 (20) | 5 (10) — Transient increases in IOP >=30 mmHg immediately following injection were collected on case report form
Dry eye (Eye disorders) | 1 (1) | 1 (2) | 2 (2)
Eyelid edema (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 3 (5) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 3 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02623426/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02623426/ICF_001.pdf